CLINICAL TRIAL: NCT05020093
Title: Clinical Performance of Injection-molded Co-cured Bulk-fill Composite Restorations Compared to Incrementally-packed Conventional Resin Composite in Proximal Cavities of Posterior Permanent Teeth: Randomized Controlled Trial
Brief Title: Clinical Performance of Injection-Molding Vs. Incremental Packing of Resin Composite in Cavitated Posterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed GS Zaghloul, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PhD2019AG
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Caries Class II
Keywords: Adhesion; Composite
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors and statistician are blinded for the type of restoration placed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection molding (Experimental): cavity design, packing technique, bonding technique
  Interventions: Procedure: Injection molding
- Incremental packing (Active Comparator): cavity design, packing technique, bonding technique
  Interventions: Procedure: Incremental packing

INTERVENTIONS:
Procedure: Injection molding — preheated bilk-fill composite, co-cured universal adhesive, David Clark cavity design
  Arms: Injection molding
Procedure: Incremental packing — Incremental packing of conventional composite; pre-cured universal adhesive, non-beveled cavity design
  Arms: Incremental packing

SUMMARY:
The clinical performance of 2 bonding and composite packing techniques in the proximal cavities of permanent posterior teeth will be assessed. Incremental packing with pre-curing of universal adhesive in selective etching mode is compared to injection molding of preheated composing co-cured with universal adhesive in selective-etch.

Main outcomes will focus on marginal integrity, post-operative hypersensitivity, and contact form and tightness.

DETAILED DESCRIPTION:
Aim of the study: To evaluate the clinical performance in terms of marginal integrity, contact tightness and form, and post-operative hypersensitivity of injection-molded co-cured bulk-fill composite versus incrementally-packed composite in proximal cavities of permanent posterior teeth.

PICOTS:

P: Population: Adult patients with carious posterior molars requiring moderate-sized proximal composite restorations I: Intervention: Injection-molding technique using co-cured bulk-fill composite resin C: Comparator: Conventional incrementally-packed resin composite O: Outcome: Primary Outcome: Marginal integrity of examined restorations; Secondary Outcomes: Post- operative hypersensitivity and contact tightness of examined restorations T: Time: Restorations will be evaluated at baseline (T0), 6 (T1), 12 (T2), 24 (T3) and 36 (T4) months. Post-operative hypersensitivity will be evaluated at 48 hours and at baseline (one week).

S: Study design: Prospective randomized controlled clinical trial (RCT): parallel, equivalence trial with 1:1 allocation ratio

Research Hypothesis:

The null hypothesis tested is that- in moderate-sized proximal cavities, there is no difference in clinical performance between injection-molded and incrementally-packed composite restorations.

Research question: In class II proximal cavities, does injection-molding of co-cured bulk-fill composites provide better clinical performance than conventional incrementally-packed composite restorations?

Study setting Study will be conducted in the Conservative Dentistry Clinic, Faculty of Dentistry- The British University in Egypt.

Interventions:

a.i. Examination and diagnosis: Examination and selection of patients will be done according to inclusion and exclusion criteria.

Upon confirming medical and dental history, recording patients' chief complaints and dentition, a pre-operative radiograph will be taken using an intraoral sensor to detect proximal caries and evaluate it against the inclusion criteria. Clinical examination will be done under 4x magnification and dental unit light using front-face dental mirror and an explorer

a.ii. Intervention:

1. Cavity preparation: Both intervention and control restorations will be placed by one operator (A.G) in a single visit per participant. Local anaesthetic agent will be administered followed by rudder dam quadrant isolation and pre-wedging using wooden wedges of appropriate sizes. Cavity preparation will be done using appropriate burs; enamel margins will be beveled, and proximal line angles will be finished using coarse and medium grit strips. Soft caries will be removed using sharp excavators of appropriate shapes and sizes. Finished cavities will be air-water rinsed to remove all blood and contaminants prior to bonding procedures.
2. Bonding procedures: Finished cavities will receive bioclear pre-contoured matrix bands of appropriate sizes. Suitable wedges and separator rings will be applied accordingly for all cavities. Etching of enamel will take place for 30 seconds with 34-37% orthophosphoric acid, which will then be rinsed off with a steady shower of air-water for 15 seconds. Cavity will be air-dried gently followed by universal adhesive application in several coats that will not be cured separately before composite injection.
3. Cavity liner: Bulk-fill flowable composite comprising 10% of the anticipated volume of the final restoration will be injected prior to the succeeding pre-heated composite paste. In this case, flowable paste is to be co-cured with the preheated successor.
4. Injection-molding procedure: a bulk-fill composite will be pre-heated in a special composite heater to 50 degrees Celsius. Composite will be dispensed from pre-heated compules into the preceding flowable paste- while maintaining the tip of the compule in the injected composite to avoid air entrapment. Both injected bulk-fill composite and preceding flowable composite will be co-cured using a LED dental lamp, checked for intensity before each procedure, according to the manufacturer's instructions.
5. Finishing and polishing: restorations will be contoured under copious coolant using medium grit diamond stones, then finished using fine-grit ones. Inter-proximal surfaces will be finished using medium and fine-grit strips. Restorations will further be polished using diamond impregnated rubber points and cups and composite polishing paste.

   1. iii. Comparator:

1- Cavity preparation: cavity preparation procedures will be carried out using appropriate rotary and hand instruments so that the final cavity will be caries free, with rounded internal line angles, saucer-shape internal outline, and finished external enamel outline. No beveling of enamel margins will take place. 2- Bonding procedures: a sectional matrix system: thin pre-contoured metal matrix of appropriate sizes, suitable wedges and separator rings will be applied to all cavities. Selective etching approach will be followed whereas enamel will be etched for 30 seconds using 34-37% orthophosphoric acid, and then rinsed off with a steady shower of air-water for 15 seconds. Cavity will be gently air dried before universal adhesive application and LED curing according to the manufacturer's instructions.

3- Cavity liner: a very thin layer of flowable composite resin will be applied over bonded surfaces, gently agitated with an explorer to clear any bubbles, then LED cured according to the manufacturer's instructions.

4- Composite resin packing: composite will be packed in a centripetal pattern using non-sticky metal composite applicators of appropriate shapes and sizes; starting with a 1 mm vertical marginal ridge followed by oblique increments, sculpted to final anatomy, and not-more-than 2 mm thick each. Each increment will be cured according to composite resin manufacturer's instruction- using a LED dental lamp checked for intensity before each procedure.

5- Finishing and polishing: restorations will be contoured under copious coolant using medium grit diamond stones, then finished using fine-grit ones. Inter-proximal surfaces will be finished using medium and fine-grit strips. Restorations will further be polished using diamond impregnated rubber points and cups and composite polishing paste.

a.iv. Assessment: Two double-blinded assessors will be calibrated to 100% agreement on 10 patients- not included in this trial. In cases of disagreement between evaluators, further discussion will take place till reaching consensus. 1ry and 2ry outcomes will be assessed following the International Dental Federation, criteria and assessment tools. Evaluation will be done at baseline (T0) (1 week after restoration); (T1) after 6 months; (T2) after 12 months; (T3) after 24 months; and (T4) at 36 months. Post-operative hypersensitivity, however, will be assessed at 48 hours and baseline only followed by vitality assessment at following recall appointments.

B. Criteria for discontinuing the intervention:

In case of pathologic or traumatic pulp injury, the process will be discontinued and the proper line of treatment will be carried out accordingly.

C. Intervention adherence:

Treatment objectives, timelines and prognosis will be explained elaborately to patients by the operator. For improving oral hygiene measures, the operator will ask the patients to adhere to oral hygiene instructions as per their follow-up instruction charts. A tooth brush and floss will be provided for each patient on each follow-up appointment.

d. Intervention-concomitant care: Patients will be instructed not to use pain killers without referring to the operator so as not to obscure the assessment of post-operative hypersensitivity.

Sample size calculation:

A success/failure response is planned to be assessed for the intended outcomes of this study- Power analysis was designed to have adequate power to apply statistical test of the research hypothesis, to evaluate bulk fill paste-like resin composite compared to conventional incremental resin composite, in restoration of carious posterior permanent teeth in terms of marginal adaptation, after 12 months using FDI criteria. According to a study in 2015, listed in the references, in which the probability of score 1 for marginal adaptation of conventional incremental resin composite (comparator) was ( 0.99); probability of score 2 was (0.01) with effect size w=0.98 (n=9). If the estimated probability of marginal adaptation for bulk fill paste-like resin composite was (0.9) for score 1, (0.1) for score 2 with effect size w= 0.8 (n=13). By adopting an alpha (α) level of 0.05 (5%), power=80%, the predicted sample size was a total of 22 (11 per group). Sample size was increased by (30%) to account for possible dropouts during follow-up intervals to be total of (28) cases i.e. (14) for each group. Sample size calculation was performed using G*Power 3.1.9.2 using chi square test.

B) Assignment of interventions:

Allocation:

a. Random sequence generation: M.Y performed block randomization; numbers were generated from 1:28 deciding which tooth to receive which intervention in each patient using online software available at www.sealedenvelope.com.

B. Allocation-concealment mechanism:

Sequence generation will be concealed using opaque sealed envelopes. Operator, A.G., will choose between numbers arranged by M.Y who will not be involved in any clinical phase.

C. Implementation: M.Y. will perform sequence concealment. A.G and M.Y will carry out allocation concealment.

Blinding (masking): It will be a triple blinded study so that subjects, assessors (A.Y and R.H), and statisticians will be blinded

C. Data collection, management and analysis a. Data collection methods:

a.i. Baseline data collection: For every patient, chief complaint, medical and dental history, and contact information will be recorded in examination charts and outpatient clinic software. Data entry will be done by A.G

1. ii. Outcome data collection: (A.Y and R.H) will be calibrated to 100% agreement on 10 patients- not included in this trial. In cases of disagreement between evaluators, further discussion will take place till reaching consensus.
2. Patient retention: A.G. will record telephone numbers and address of all subjects in the study as a part of the signed consent. Patients will be contacted by phone one day before the follow-up dates. A.G will also explain to the patient the benefits of follow up and any defective restoration will be managed accordingly.

Data management:

A.G will electronically enter all the data. Patients' files are to be stored in numerical order in a secured place. All paper sheets concerned with the personal or outcome data will be stored in a locked cabinet and the Conservative dentistry department, the British University in Egypt. The excel sheets of patients data will be stored in a computer in the Conservative Department- Faculty of Dentistry, the British University in Egypt. The computer will have a password only known to A.G and M.Y. to prevent unauthorized access to data and double data entry. A back-up will be made online to avoid data loss.

Statistical methods:

Qualitative data will be presented as percentages. Chi-square test or Fisher's exact test when applicable will be used for comparisons between the groups. Friedman's test and Kaplan-Meier plot will be used to study the changes by time. Log-rank test will be used to statistically compare the groups when evaluating survival analysis. The significance level will be set at P ≤ 0.05. Statistical analysis will be performed with IBM® SPSS® Statistics Version 20 for Windows (SPSS, Inc., an IBM Company).

D. Data monitoring:

Monitoring:

M.Y will monitor this study for the risk of bias and to monitor blinding. She will also have full access to the results and to take the final decision to terminate the trial when necessary.

Harms:

A.G will explain possible harms to patients. o harms are expected and if the is any adverse actions, the process will be stopped immediately and managed accordingly after reporting it to M.Y and R.H.

Auditing:

Auditing of the study design will be done by M.Y and R.H the co-supervisor to assure quality of the research procedures

ELIGIBILITY:
Inclusion Criteria:

- Patients with a minimum of one proximal carious lesion in a maxillary or mandibular posterior tooth

* Selected teeth should have not more than one proximal carious lesion
* Caries should be extending not more than the outer third of dentin in pre-operative radiograph
* Presence of antagonist and adjacent teeth for selected molars
* Vital teeth with no signs or symptoms of pulpitis
* Anticipated cavity external walls should be in enamel
* Normal periodontal status and good oral hygiene
* Mobility grade ≤ 1
* Good general health

Exclusion Criteria:

* Patients with occlusal, buccal or lingual caries lesions in selected teeth

  * Two proximal cavities in selected teeth
  * Extensive carious lesions; shallow enamel lesions or old restorations
  * Absence of antagonist or adjacent teeth
  * Non-vital, hyperemic or endo-treated teeth
  * Cavities requiring gingival margin relocation or pulp capping (direct or indirect)
  * Chronic or acute periodontitis
  * Mobility grade 2 or 3
  * >50 and <18 Years old
  * Systemic conditions, allergy to restorative materials and hospitalized patients
  * Evidence of bruxism and temporomandibular joint disorders
  * Patients with low compliance potential

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Marginal integrity using a 150- and 250- micron width special probe tip | 36 months
  gap width at tooth-restoration interface

SECONDARY OUTCOMES:
Post-Operative hypersensitivity: using Visual Analog Scale 0-10 (VAS). Zero: no pain; 10: unbearable pain. | 48 hours and one week
  post-operative reported pain
Contact tightness: gap width between proximal teeth surfaces. Using a 25-micron dental floss, and 50- and 100- micron metal blade | 36 months
  Contact tightness and proximal surface form

CONTACTS AND LOCATIONS:
Overall Officials: Randa Mohamed, Study Chair — Professor of Conservative Dentistry
Locations (1):
- The British university in Egypt, Cairo, Egypt

REFERENCES:
- [Result] Kitasako Y, Sadr A, Burrow MF, Tagami J. Thirty-six month clinical evaluation of a highly filled flowable composite for direct posterior restorations. Aust Dent J. 2016 Sep;61(3):366-73. doi: 10.1111/adj.12387. PMID 26573239